CLINICAL TRIAL: NCT00750503
Title: Workplace Tobacco Cessation And Oral Cancer Screening Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tata Memorial Hospital (Other Government)
Collaborators: Department of Atomic Energy (Other Government)
Responsible Party: Dr. Gauravi Ashish Mishra, Assistant Professor and Assistant Physician, Tata Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 458
Record Dates: First submitted 2008-09-09; First posted 2008-09-10 (Estimated); Last update posted 2008-09-10 (Estimated); Status verified 2008-08

CONDITIONS: Tobacco Cessation; Oral Cancer
Keywords: tobacco cessation; behavioral therapy; pharmacotherapy; workplace; oral cancer screening; Tobacco Quit rates
MeSH Terms: conditions — Tobacco Use Cessation; Mouth Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Behavioural and Pharmacotherapy for tobacco cessation — Professional help in the form of health awareness sessions, focus group discussion, one to one counseling and pharmacotherapy was provided to the employees by a team of doctors and counselors from Tata Memorial Hospital. Self reporting of tobacco history was validated with Rapid Urine cotinine test. Naked eye examination of oral cavity of all employees for detection of oral pre-cancers and cancers was conducted. Nursing staff and Doctors attached to the industry and from the local referral hospital were invited to participate as trainees during the active intervention sessions for local manpower development.

SUMMARY:
Tata Memorial Hospital has initiated Workplace Tobacco Cessation and Oral Cancer Screening Programme in Chemical Industry at Khed, Ratnagiri. Appropriate interventions for tobacco cessation will be carried at monthly intervals for twelve months duration. The tobacco cessation rates based on history will be validated with the urinary cotinine levels.

DETAILED DESCRIPTION:
The prevalence of tobacco use in India among men has been reported to be high in most parts (generally exceeding 50%). It's use is more common in rural areas as compared to urban areas. Oral cancer, the main cause of which is tobacco, is common in men in developing countries and the most common cancer among men in India. The five year survival rate for oral and pharyngeal cancers even in premier institute like the Tata Memorial Hospital ranges from a poor 8% (hypo pharynx) to 43% (lower lip). Evidence has shown that cessation is the only intervention with the potential to reduce tobacco related mortality in the short- term and medium- term. An emphasis on prevention of tobacco consumption will, in the short run, only have a limited positive effect on tobacco related morbidity and mortality, as prevention strategies do not affect existing consumers. Workplace tobacco cessation activities in India are still in rudimentary stage.

In the proposed study of one year duration, professional help in the form focus group discussion, one to one counseling and pharmacotherapy will be provided to the employees by a team of doctors and counsellors from Tata Memorial Hospital. Self reporting of tobacco history will be validated with Biochemical test. This will add objectivity to the programme, so that, if successful, it can be replicated as a model to promote tobacco control activities at other workplaces. Naked eye examination of oral cavity of all employees for detection of oral pre-cancers and cancers will be done by doctors from the Tata Memorial Hospital. The employees with lesions may be referred for further management, if required. Nursing staff and Doctors attached to the industry and from the local referral hospital will be invited to participate as trainees during the active intervention sessions.

The long term objective of this initiative is to establish a model workplace tobacco cessation and oral cancer screening programme. It will contribute to the human resource and infrastructure development for tobacco cessation services at the industrial unit and at the local referral hospital. Proposed tobacco cessation services in the chemical industry would be of great help for boosting Anti - Tobacco Activities not only in the particular factory unit but also in the nearby industrial and residential zone.

ELIGIBILITY:
Inclusion Criteria:

* All 104 employees working in the chemical industrial unit at Khed, Ratnagiri, are eligible to participate.

Exclusion Criteria:

* There are no exclusion criteria.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2007-06; Primary Completion 2008-06 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
The prevalence of tobacco use and the the change in Knowledge, Attitude and Practices during post intervention. The reasons for initiation and continuation of tobacco consumption habit. The tobacco quit rates. | 12 months

SECONDARY OUTCOMES:
The prevalence of oral precancerous and cancerous lesions among this group and its correlation with the different forms and frequency of tobacco use. | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Chemical Industry, Tal. Khed, District : Ratnagiri, Maharashtra, India